CLINICAL TRIAL: NCT00401986
Title: Long Term Safety Evaluation of Bronchial Thermoplasty With the Alair® System in Patients With Severe Asthma
Brief Title: RISA Extension Study - Long Term Safety
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 06-01
Record Dates: First submitted 2006-11-17; First posted 2006-11-22 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Refractory Asthma; Bronchial Thermoplasty; Alair System; RISA (Research in Severe Asthma)
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Alair Treatment: Alair Treated subjects from PREDECESSOR STUDY (NCT00214539).
  Interventions: Device: Bronchial thermoplasty with the Alair System

INTERVENTIONS:
Device: Bronchial thermoplasty with the Alair System — Treatment of airways with the Alair System in PREDECESSOR STUDY (NCT00214539).

SUMMARY:
The primary purpose of this study is to gather additional safety data for the subjects treated with the Alair System (hereinafter, "Alair-Treated Subjects") who previously completed the one-year study entitled: "Multicenter Randomized Clinical Trial of Bronchial Thermoplasty with the Alair System for the Treatment of Severe Asthma" (Protocol #0903-27) sponsored by Asthmatx, Inc. Subjects who elect to participate in this safety study will be followed for an additional four (4) year period beyond the PREDECESSOR STUDY'S one-year endpoint (clinicaltrials.gov number NCT00214539).

DETAILED DESCRIPTION:
This will be a multicenter study conducted only at the clinical sites that participated in the PREDECESSOR STUDY (NCT00214539).

Enrollment will be limited to only those subjects who were treated with the Alair System in the PREDECESSOR STUDY.

Written, informed consent will be obtained from all subjects prior to performing any study procedures.

The present study will extend the follow-up evaluation of Alair-Treated Subjects from the PREDECESSOR STUDY to 5 years post-treatment with the Alair System. These evaluations will consist of four study visits corresponding to the two-year, three-year, four-year and five-year time points following completion of Alair treatments in the PREDECESSOR STUDY. For consistency with the PREDECESSOR STUDY, ideally the subject's drug therapy should continue to be consistent with GINA (Global Initiative for Asthma) Guidelines for the severity of the subject's asthma. Any changes in maintenance levels of asthma medications will be documented.

The goal of this follow-on study is to enroll all Alair-Treated Subjects who completed the PREDECESSOR STUDY. Inclusion of subjects from the treatment arm will allow for better assessment of the long-term safety of the Alair procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subject who participated in the PREDECESSOR STUDY entitled "Multicenter Randomized Clinical Trial of Bronchial Thermoplasty with the Alair™ System for the Treatment of Severe Asthma" (Protocol # 0903-27).
* Subject was treated with the Alair System ("Alair Group") in the PREDECESSOR STUDY.
* Subject who is able to read, understand, and provide written Informed Consent.
* Subject who is able to comply with the study protocol, including requirements for taking and abstaining from medications, and complete all study required visits.

Exclusion Criteria:

* Subject participating in another clinical trial involving respiratory intervention that could affect the outcome measures of this study, either within 6 weeks of study enrollment, or during the study period.
* Subject with a newly diagnosed (since exiting from the PREDECESSOR STUDY) psychiatric disorder which in the judgment of the investigator could interfere with provision of informed consent, completion of tests, therapy, or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with severe asthma, previously treated with the Alair System in the PREDECESSOR STUDY (NCT00214539).
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder S Shargill, PhD, Study Director — Asthmatx, Inc.
Locations (8):
- Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (2):
  - St. Joseph's Healthcare, Hamilton, Ontario
  - Hospital Laval, University of Laval, Sainte-Foy, Quebec
- United Kingdom (5):
  - Gartnavel General Hospital, Univ. Glasgow, Glasgow
  - Glenfield General Hospital, Univ. Leicester, Leicester
  - National Heart and Lung Institute, Imperial College, London
  - Northwest Lung Research Center, University of Manchester, Manchester
  - William Leech Center, Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pavord ID, Cox G, Thomson NC, Rubin AS, Corris PA, Niven RM, Chung KF, Laviolette M; RISA Trial Study Group. Safety and efficacy of bronchial thermoplasty in symptomatic, severe asthma. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1185-91. doi: 10.1164/rccm.200704-571OC. Epub 2007 Sep 27. PMID 17901415
- [Background] Thomson NC, Rubin AS, Niven RM, Corris PA, Siersted HC, Olivenstein R, Pavord ID, McCormack D, Laviolette M, Shargill NS, Cox G; AIR Trial Study Group. Long-term (5 year) safety of bronchial thermoplasty: Asthma Intervention Research (AIR) trial. BMC Pulm Med. 2011 Feb 11;11:8. doi: 10.1186/1471-2466-11-8. PMID 21314924
- [Result] Pavord ID, Thomson NC, Niven RM, Corris PA, Chung KF, Cox G, Armstrong B, Shargill NS, Laviolette M; Research in Severe Asthma Trial Study Group. Safety of bronchial thermoplasty in patients with severe refractory asthma. Ann Allergy Asthma Immunol. 2013 Nov;111(5):402-7. doi: 10.1016/j.anai.2013.05.002. Epub 2013 Jun 13. PMID 24125149

RESULTS

PARTICIPANT FLOW:
Groups:
- Alair Group: A total of 14 Alair group subjects from the PREDECESSOR STUDY (NCT00214539) provided consent and participated in the RISA Extension Study evaluating the longer-term safety of the Alair treatment.
Period: Overall Study
Arm/Group | Alair Group
Started | 14
Completed | 12
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Alair Group: Baseline Demographics are based on data collected at the time of entry into the PREDECESSOR STUDY (NCT00214539).
Arm/Group | Alair Group
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.64 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 4
  United Kingdom | 10
amPEF (Peak Expiratory Flow) [Mean (Standard Deviation); unit: L/min (liters per minute)] | 369.95 (82.04)
Pre-Bronchodilator FEV1 (Forced Expiratory Volume in 1 second) [Mean (Standard Deviation); unit: % predicted] | 63.46 (12.49)
Post-Bronchodilator FEV1 [Mean (Standard Deviation); unit: % predicted] | 75.19 (11.91)
ICS Dose (Inhaled Corticosteroid dose) [Mean (Standard Deviation); unit: µg/day (microgram/day)] | 1179 (421)
LABA Dose (Long-acting Beta Agonists) [Mean (Standard Deviation); unit: µg/day (microgram/day)] | 127 (62)
OCS Dose (Oral corticosteroids) [Mean (Standard Deviation); unit: mg/day (milligrams/day)] | 13.6 (6.3)
Rescue Medication Use [Mean (Standard Deviation); unit: Puffs/7 days] | 60.9 (60.9)
Asthma Control Questionnaire (ACQ) Score [Mean (Standard Deviation); unit: scores on a scale] — The ACQ has 7 questions (the top scoring 5 symptoms, FEV1% predicted and daily rescue bronchodilator use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). Clinic staff score the FEV1% predicted on a 7-point scale. The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled).
  scores on a scale | 2.76 (1.02)
Asthma Quality of Life Questionnaire (AQLQ) Score [Mean (Standard Deviation); unit: scores on a scale] — There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains.
  scores on a scale | 4.11 (1.27)
Symptom-Free Days [Mean (Standard Deviation); unit: percentage of days] — Symptom-Free Days were defined as days when Subject reported no cough, wheeze, breathlessness, or sputum during the daytime, and no wheeze, cough, or awakenings due to asthma symptoms during nighttime.
  percentage of days | 5.61 (14.06)
Total Symptom Score [Mean (Standard Deviation); unit: scores on a scale] — Total Symptom Score comprises the sum of these six asthma symptom measurements: wheeze during the night, cough during the night, wheeze during the day, cough during the day, breathlessness during the day, and sputum production during the day. Each of these symptoms is scored on a scale of 0 to 3 each day by the subject. The sum of the scores for these 6 symptoms comprises the Total Symptom Score, which measures overall asthma symptoms. The maximum score possible is 18; the minimum possible score is 0. A lower Total Symptom score represents better asthma control.
  scores on a scale | 5.35 (2.92)
Unscheduled Physician Office Visits [Number; unit: Number of events] — Number of Events (number of Subjects) = 8 (6)
  Number of events | 8
Emergency Room Visits [Number; unit: Number of events] — Number of Events (number of Subjects) = 5 (4)
  Number of events | 4
Hospitalizations [Number; unit: Number of events] — Number of Events (number of Subjects) = 10 (6)
  Number of events | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Respiratory Adverse Events (AEs) in Annual Increments
Description: The respiratory-related adverse event profile for the Alair group was analyzed on an annual basis in order to highlight trends in adverse occurrence.
Time Frame: 2-year, 3-year, 4-year and 5-year follow up post procedure
Population: A total of 14 Alair group subjects from the PREDECESSOR STUDY (NCT00214539) provided consent and participated in the RISA Extension Study evaluating the longer-term safety of the Alair treatment. All 14 subjects completed their Year 3 visit and 12 subjects have completed their Year 4 and 5 visits.
Measure: Number; unit: percentage subjects with respiratory AEs
Groups:
- Alair Group: A total of 14 Alair group subjects from the PREDECESSOR STUDY (NCT00214539) provided consent and participated in the RISA Extension Study evaluating the longer-term safety of the Alair treatment.
  A total of 145 adverse events have been reported by the 14 subjects enrolled in the present study over Year 2 through 5. One hundred and three adverse events (71%) were respiratory-related.
  The number of subjects reporting respiratory-related adverse events each year was consistent. Reporting were 11/14 subjects (78.6%) in Year 2, 12/14 subjects (85.7%) in Year 3, 10/12 subjects (83.3%) in Year 4, and 12/12 subjects (100%) in Year 5 reported respiratory adverse events.
Arm/Group | Alair Group
Number analyzed (Participants) | 14
percentage subjects with respiratory AEs
  Year 2, n=14 | 78.6
  Year 3, n=14 | 85.7
  Year 4, n=12: number analyzed (Participants) | 12
  Year 4, n=12 | 83.3
  Year 5, n=12: number analyzed (Participants) | 12
  Year 5, n=12 | 100

2. Primary Outcome: Respiratory Adverse Events
Description: Pull down menu does not have a rate unit. Numbers reported represents Rate of Respiratory Adverse (number of Events/number of Subject/year).
Time Frame: 2-year, 3-year, 4-year and 5-year follow up post procedure
Population: Subject attrition at years 4 & 5
Measure: Number; unit: Number of events/number of subject/Year
Arm/Group | Alair Group
Number analyzed (Participants) | 14
Number of events/number of subject/Year
  Year 2, n=14 | 1.4
  Year 3, n=14 | 2.4
  Year 4, n=12: number analyzed (Participants) | 12
  Year 4, n=12 | 1.7
  Year 5, n=12: number analyzed (Participants) | 12
  Year 5, n=12 | 2.4

3. Secondary Outcome: Hospitalizations for Respiratory Symptoms
Description: Pull down menu does not have a rate unit. Rate of Hospitalizations for Respiratory Symptoms (number of Events/number of Subject/year)
Time Frame: 2-year, 3-year, 4-year and 5-year follow up post procedure
Population: Subject attrition at years 4 & 5
Measure: Number; unit: Number of events/number of subject/Year
Groups:
- Alair Group: A total of 14 Alair group subjects from the PREDECESSOR STUDY (NCT00214539) provided consent and participated in the RISA Extension Study evaluating the longer-term safety of the Alair treatment.
  .
Arm/Group | Alair Group
Number analyzed (Participants) | 14
Number of events/number of subject/Year
  Year 2, n=14 | 0.4
  Year 3, n=14 | 0.2
  Year 4, n=12: number analyzed (Participants) | 12
  Year 4, n=12 | 0.1
  Year 5, n=12: number analyzed (Participants) | 12
  Year 5, n=12 | 0.1

4. Secondary Outcome: Emergency Room Visits for Respiratory Symptoms
Description: Pull down menu does not have a rate unit. Rate of Emergency Room Visits for Respiratory Symptoms (number of Events/number of Subjects/year)
Time Frame: 2-year, 3-year, 4-year and 5-year follow up post procedure
Population: Subject attrition at years 4 & 5
Measure: Number; unit: Number of events/number of subject/Year
Arm/Group | Alair Group
Number analyzed (Participants) | 14
Number of events/number of subject/Year
  Year 2, n=14 | 0.3
  Year 3, n=14 | 0
  Year 4, n=12: number analyzed (Participants) | 12
  Year 4, n=12 | 0
  Year 5, n=12: number analyzed (Participants) | 12
  Year 5, n=12 | 0.1

ADVERSE EVENTS:
Time Frame: Year 2 post procedure out to 5 years (total of 4 years). 14 Alair group subjects from the PREDECESSOR STUDY (NCT00214539) participated in the RISA Extension Study.
Groups:
- Year 2; Year 3; Year 4; Year 5: Conventional therapy with high dose ICS+LABA±OCS (≤30mg/day) plus Alair Treatment
Arm/Group | Year 2 | Year 3 | Year 4 | Year 5
Serious Adverse Events (participants affected / at risk) | 5/14 | 4/14 | 3/12 | 3/12
Other Adverse Events (participants affected / at risk) | 11/14 | 12/14 | 11/12 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 2 (N=14) | Year 3 (N=14) | Year 4 (N=12) | Year 5 (N=12)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Respiratory
Sudden Death (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) — Non-Respiratory
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 0 (0) | 1 (1) — Respiratory
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Respiratory
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Nocturnal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory
Asthma exacerbation prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Respiratory
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 2 (N=14) | Year 3 (N=14) | Year 4 (N=12) | Year 5 (N=12)
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 (11) | 7 (12) | 2 (3) | 4 (4) — Respiratory
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4) | 1 (1) | 1 (1) — Respiratory
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Respiratory
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) — Respiratory
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Respiratory
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5) | 5 (8) | 7 (11) — Respiratory
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Respiratory
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) — Respiratory
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Respiratory
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Respiratory
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Respiratory
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (3) | 2 (3) — Respiratory
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) — Respiratory
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Respiratory
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Respiratory
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Respiratory
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Venipuncture site thrombosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Gastroenteritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Respiratory
Whiplash injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Respiratory
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) — Non-Respiratory
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Non-Respiratory
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-Respiratory
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Respiratory
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-Respiratory
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-Respiratory
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Non-Respiratory
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-Respiratory
Asthma exacerbation prophylaxis (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Non-Respiratory

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less